CLINICAL TRIAL: NCT07184866
Title: A Randomized Controlled Trial Open Label Evaluating the Efficacy of Vitamin C in Improving Outcomes of Acute Kidney Injury in Patients With ACLF With Septic Shock
Brief Title: Vitamin C for Acute Kidney Injury in ACLF With Septic Shock: A Randomized Controlled Trial
Acronym: VITAKI-ACLF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Principal Investigator, Rakhi Maiwall, Professor (hepatology), Institute of Liver and Biliary Sciences, India
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IEC/2024/116/MA02; IEC approval number (Other: Institute of Liver and Biliary Sciences)
Record Dates: First submitted 2025-09-13; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Acute-on-Chronic Liver Failure (ACLF)
Keywords: Sepsis, septic shock, Alcohol-related, ACLF, AKI, Lactate, Vitamin
MeSH Terms: conditions — Acute-On-Chronic Liver Failure; Sepsis; Shock, Septic | interventions — Ascorbic Acid; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (SOC) (Active Comparator): Participants in this arm will receive standard medical treatment for ACLF with septic shock and acute kidney injury, as per institutional protocols.
  Interventions: Other: Standard of Care (SOC)
- Vitamin C + Standard of Care (Experimental): Participants in this arm will receive intravenous Vitamin C (25 mg/kg, up to 1.5 g every 6 hours for 5 days) in addition to standard medical treatment for ACLF with septic shock and acute kidney injury
  Interventions: Drug: Vitamin C

INTERVENTIONS:
Drug: Vitamin C — Intravenous Vitamin C, 25 mg/kg (maximum 1.5 g) every 6 hours for 5 days, administered in addition to standard medical treatment
  Other Names: (Ascorbic Acid)
  Arms: Vitamin C + Standard of Care
Other: Standard of Care (SOC) — Supportive and guideline-based management of ACLF with septic shock and AKI, including antibiotics, fluids, vasopressors, renal replacement therapy as required, and other standard therapies
  Arms: Standard of Care (SOC)

SUMMARY:
This study is testing whether Vitamin C can help improve kidney function and survival in very sick patients with liver disease. Patients with acute-on-chronic liver failure (ACLF) often develop serious infections that can lead to septic shock and kidney injury, which are major causes of death.

In this randomized controlled trial, patients with ACLF and septic shock will be assigned to receive either:

1. Standard medical treatment alone, or
2. Standard medical treatment plus intravenous Vitamin C.

Vitamin C is a safe, inexpensive antioxidant that may reduce inflammation, improve circulation, and protect the kidneys. The study will compare how well patients recover from septic shock and kidney injury in the two groups. Blood and urine samples will also be collected to look for biological markers that can predict outcomes.

DETAILED DESCRIPTION:
Acute-on-chronic liver failure (ACLF) is a severe condition in which patients with chronic liver disease suddenly develop liver failure, often triggered by infection. Many of these patients progress to septic shock, and acute kidney injury (AKI) is a common and life-threatening complication. Current treatment options are limited, and mortality remains very high.

Vitamin C is a low-cost, widely available antioxidant and immune-modulating agent. It has shown promising results in patients with sepsis and septic shock by reducing oxidative stress, improving vascular tone, and supporting immune defense. However, its role in ACLF patients with septic shock and AKI has not been studied in a large, controlled trial.

This interventional, randomized, open-label controlled trial will enroll patients with alcohol-related ACLF, septic shock, and AKI. Participants will be randomized 1:1 to receive either intravenous Vitamin C in addition to standard medical care, or standard care alone. Clinical outcomes, including resolution of shock, progression or resolution of AKI, need for renal replacement therapy, ICU/hospital stay, and survival at 7 and 28 days will be assessed. In addition, biospecimens (blood and urine) will be analyzed to identify biomarkers that predict outcomes and response to Vitamin C therapy.

The study aims to provide evidence on the effectiveness of Vitamin C as an adjunctive therapy in this high-risk population, and to generate insights into the mechanisms of septic shock and kidney injury in ACLF.

ELIGIBILITY:
Inclusion Criteria:

* ACLF as per asia pacific association for the study of liver (APASL criteria) with AKI according to KDIGO Criteria and septic shock.

Exclusion Criteria:

* • Refractory Septic shock with more than 3 organ failures.

  * Patients with age less than 18 years
  * Known severe cardiopulmonary disease (structural or valvular heart disease, coronary artery disease, COPD)
  * Patients in DIC with platelets < 20,000 and INR > 4 or active bleeding
  * Limitations of care (defined as refusal of cardiovascular and respiratory support modes) including "do not intubate" (DNI) status
  * Current hospitalization > 15 days for patients with nosocomial acquisition of MDR at time of randomization
  * Known allergy or contraindication to vitamin C (including previously or currently diagnosed primary hyperoxaluria and/or oxalate nephropathy, or known/suspected ethylene glycol ingestion,
  * Known glucose-6-phosphate dehydrogenase (G6PD) deficiency)
  * Use of vitamin C at a dose of > 1 gram daily within the 24 hours preceding first episode of qualifying organ dysfunction during a given ED or ICU admission
  * Patients with HCC (beyond Milan) or extrahepatic malignancies
  * Patients with HVOTO or EHPVO
  * Pregnancy or active breastfeeding
  * Current participation in another interventional research study
  * Active or history of kidney stones
  * History of chronic kidney disease or intrinsic kidney disease
  * Patients already on maintenance hemodialysis prior to presentation
  * Failure to provide informed consent
  * Patients with retroviral infection
  * Patients with active hemolysis due to alcohol or other causes or with hemoglobin below 7 gm/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Resolution of septic shock at 96 hours (Day 4) | Day 4 (96 hours) after randomization
  Resolution of septic shock is defined as maintenance of mean arterial pressure (MAP) ≥ 65 mmHg for ≥ 6 consecutive hours after complete discontinuation of all vasopressor support, without restarting vasopressors during that 6-hour period.

SECONDARY OUTCOMES:
Outcome of acute kidney injury (AKI) at Day 7 | Day 7
  AKI resolution (decrease in stage by ≥1 or return to no AKI), persistence (same stage), or progression (increase in stage by ≥1 or need for dialysis in stage 3 patients), defined by KDIGO criteria.
Incidence of adverse events | Day 7, Day 14, Day 28 or until hospital discharge, whichever occurs first
  Number and type of adverse events including hypotension, sepsis, bleeding, allergic reactions, anemia, kidney stones, urinary oxalate, hemolysis, and thrombocytopenia.
Need for renal replacement therapy | Day 7
  Proportion of patients requiring initiation of renal replacement therapy.
Duration of ICU stay | Through hospital discharge or death, up to 28 days
  Number of days spent in ICU from randomization to discharge or death.
Duration of hospital stay | Up to Day 28
  Total number of days from admission to discharge or death.
7-day mortality | Day 7
  All-cause mortality within 7 days of randomization
28-day mortality | Day 28
  All-cause mortality within 28 days of randomization